CLINICAL TRIAL: NCT02694172
Title: Analysis of the Diversity of Faecal Bacteria in Healthy and Type 2 Diabetic Subjects
Brief Title: Human Faecal Microbiota in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University Hospital, Geneva (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06.42.NRC
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes; Healthy; Overweight
Keywords: diabetes mellitus type 2; healthy subjects; human microbiome; cereal bar
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lean non diabetic (No Intervention): Lean and healthy subjects receiving no intervention
- Overweight non diabetic (Experimental): fiber rich cereal bars, two bars a day for 4 weeks
  Interventions: Other: Fiber rich cereal bars
- Overweight diabetic (Experimental): fiber rich cereal bars, two bars a day for 4 weeks
  Interventions: Other: Fiber rich cereal bars

INTERVENTIONS:
Other: Fiber rich cereal bars — Two cereals per day and per subject for 4 weeks
  Other Names: Nutren balance bars
  Arms: Overweight diabetic; Overweight non diabetic

SUMMARY:
The main objective of the clinical trial is to investigate whether overweight type 2 diabetic patients have a different fecal microbiota profile compared with age, gender, BMI matched subjects and with lean healthy subjects before and after the consumption of fiber rich cereal bars.

DETAILED DESCRIPTION:
Gut microbiota refers to the bacterial communities in the gastrointestinal tract. The diversity and quantity of bacteria vary depending on age of the individuals, daily diet and the segment of the intestine, which makes the gut microbiota one of the most complex bacterial ecosystems known to men. In general, over trillions of bacteria reside in human gut. Recent evidence indicates that gut microbiota could be involved in host metabolism by multiple pathways leading to the development of obesity and type 2 diabetes. Increased fat storage or obesity has become one of the leading public health issues in many developed and developing countries. However, it is not clear whether type 2 diabetes is associated with a unique gut microbiota profile. Therefore, the primary objective of the study is to compare the fecal microbiota of overweight type 2 diabetic subjects to that of age, gender and BMI matched subjects as well as with lean non-diabetic subjects. In addition, the investigators hypothesize that microbiota modifications with consumption of fiber rich food products can improve the metabolic outcomes of type 2 diabetics. To test this hypothesis, the investigators plan to provide each overweight participant with two cereal bars per day for 4 weeks. Anthropometric measurements and plasma parameters as well as the fecal microbiota will be determined.

ELIGIBILITY:
Inclusion Criteria:

-All diabetic and control non-diabetic subjects (of same BMI) must comply with all the following inclusion criteria:

* Ethnic background: Caucasian
* BMI: 25 to 40 kg/m2
* Fasting blood glucose > 7 mmol/L
* Fasting Hemoglobin A1c > 7%
* Consume mainly typical Western diets daily
* Having obtained his/her informed consent

Lean non-diabetic healthy subjects must comply with the following inclusion criteria:

* Ethnic background: Caucasian
* BMI: 20 to 25 kg/m2
* Fasting blood glucose < 5.5 mmol/L
* Fasting Hemoglobin A1c < 6 %
* Consume mainly typical Western diets daily
* Having obtained his/her informed consent

Exclusion Criteria:

Diabetic and healthy (same BMI) subjects representing one or more of the following criteria are excluded from participation in the study.

* Dietary supplements or medications known to alter gut bacteria, such as antibiotic medication or intestinal transit modulators
* People actively take cortisol or dexamethasone should be excluded from the study
* People under a-amylase/a-glucosidase inhibitors should be excluded from the study. However, patients under metformin can be accepted for this study.
* Patients under metformin suffering from gastrointestinal side effects within a 6-month time period prior to the trial
* Regular consumption of fermented dairy products
* Vegetarians
* Frequent diarrhea (more than two loose stool per day) within 7 days before the enrollment
* HIV seropositive
* Having known gastrointestinal diseases such as ulcerative colitis, Crohn's disease, peptic ulcers and cancer
* Patients who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 6 months prior to the beginning of this study
* Females with hormone therapy will be excluded from the study

Lean healthy subjects representing one or more of the following criteria are excluded from participation in the study.

* Dietary supplements or medications known to alter gut bacteria, such as antibiotic medication or intestinal transit modulators
* Regular consumption of fermented dairy products
* Vegetarians
* Frequent diarrhea (more than two loose stool per day) within 7 days before the enrollment
* HIV seropositive
* Having known gastrointestinal diseases such as ulcerative colitis, Crohn's disease, peptic ulcers and cancer
* Patients who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 6 months prior to the beginning of this study
* Females with hormone therapy will be excluded from the study

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota profile | Baseline samples taken after 2 weeks of diet normalization period
  Fecal samples taken after the two week diet normalization are subjected to bacteria 16S rDNA sequencing and by quantitative PCR.

SECONDARY OUTCOMES:
Metabonomic analysis in faeces | Samples taken after 2 weeks of diet normalization period (baseline) and 4 weeks of cereal bars intake when applicable
  Samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects. Then, samples are analyzed by 1HNMR.
Metabonomic analysis in plasma | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects. Then, samples are analyzed by 1HNMR.
Metabonomic analysis in urine | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects. Then, samples are analyzed by 1HNMR.
Plasma glucose | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.
Plasma insulin | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.
Plasma free fatty acids | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.
Plasma triglycerides | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.
Plasma total cholesterol | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.
Plasma HDL cholesterol | Samples taken after 2 weeks of diet normalization period and 4 weeks of cereal bars intake when applicable
  Baseline samples for lean non-diabetic, overweight non-diabetic and overweight diabetic subjects. Post intervention samples from overweight non-diabetic and diabetic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Golay, Prof, Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: No